CLINICAL TRIAL: NCT01237795
Title: A Randomized Trial of Experimental Dentifrices for Cleaning Dentures
Brief Title: Experimental Denture Pastes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raphael Freitas de Souza (Other)
Responsible Party: Sponsor-Investigator, Raphael Freitas de Souza, Associate Professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FORP-PT-003; 2008.1.33.58.7 (Other: Institutional Review Board (FORP-USP))
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Dental Plaque; Denture Stomatitis; Oral Candidiasis; Oral Hygiene
Keywords: Chloramine T; Complete Denture; Dental Plaque Index; Dentifrice; Denture Bases; Denture Cleansers; Edentulous Mouth; Fluorosurfactant; Oral Health; Toothpaste
MeSH Terms: conditions — Dental Plaque; Stomatitis, Denture; Candidiasis, Oral; Mouth, Edentulous | interventions — Dentifrices; Toothpastes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.01% fluorosurfactant (Experimental): An experimental formula for denture hygiene containing 0.01% fluorosurfactant.
  Interventions: Other: Dentifrice
- 1.0% chloramine T (Experimental): An experimental formula for denture hygiene containing 1.0% chloramine T.
  Interventions: Other: Dentifrice
- 0.2% chloramine T (Experimental): An experimental formula for denture hygiene containing 0.2% chloramine T.
  Interventions: Other: Dentifrice
- Proprietary dentifrice. (Active Comparator): A proprietary denture-specific dentifrice.
  Interventions: Other: Dentifrice

INTERVENTIONS:
Other: Dentifrice — Dentifrices (4 formulations) used as auxiliary agents for brushing complete dentures.
  Other Names: Denture-specific paste; Toothpaste

SUMMARY:
This trial aims to evaluate the efficacy of three experimental dentifrices to remove denture biofilm. Complete denture wearers will be instructed to brush their dentures with a specific toothbrush and four compositions: (1) A proprietary denture-specific paste (active comparator); (2) 0.2% chloramine T; (3) 1.0% chloramine T; (4) 0.01% fluorosurfactant. Each treatment will be used for periods of 7 days, and participants will be randomized to use them according to one of four sequences.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous
* Good general health
* Patients requesting new complete dentures (volunteers will receive the interventions before new complete dentures)
* Regular wearing of the same maxillary and mandibular complete dentures for 3 to 10 years
* Both denture bases and artificial teeth should be composed by acrylic resin

Exclusion Criteria:

* Unsatisfactory complete dentures in use (i.e. with poor fitting, relining or fractures)
* Absence of deposits of biofilm at baseline

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Denture plaque coverage area (%) | 7 days
  Relation between stained area and total surface area on the internal surface of maxillary complete dentures.

CONTACTS AND LOCATIONS:
Overall Officials: Helena FO Paranhos, DDS, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Ribeirão Preto Dental School, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Institutional page of the Ribeirão Preto Dental School (research site) — http://www.forp.usp.br
- See also: Principal Investigator´s CV — http://lattes.cnpq.br/6275169074451249